CLINICAL TRIAL: NCT00639743
Title: Comparison Trial Evaluating Efficacy and Safety of Single i.v. Bolus Tenecteplase Plus Standard Anticoagulation as Compared With Standard Anticoagulation in Normotensive Patients
Brief Title: PEITHO Pulmonary Embolism Thrombolysis Study
Acronym: PEITHO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government); Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P030444
Record Dates: First submitted 2008-03-13; First posted 2008-03-20 (Estimated); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Pulmonary Embolism
Keywords: Pulmonary embolism; Heparin; Thrombolytic therapy; Bleeding
MeSH Terms: conditions — Pulmonary Embolism; Hemorrhage | interventions — Tenecteplase

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- group A (Experimental): tenecteplase (group A)
  Interventions: Drug: tenecteplase (group A)
- group B (Placebo Comparator): placebo ( group B)
  Interventions: Drug: placebo ( group B)

INTERVENTIONS:
Drug: placebo ( group B) — placebo ( group B)
  Arms: group B
Drug: tenecteplase (group A) — tenecteplase (group A)
  Arms: group A

SUMMARY:
Heparin is the reference therapy for most patients with pulmonary embolism. Some patients with sub-massive pulmonary embolism defined by normal blood pressure and dysfunction of the right ventricle have a higher mortality risk. It has been suggested that thrombolytic treatment, a drug that dissolves blood clots more rapidly, may reduce the mortality in those patients. The studies reported to date were unable to confirm or refute this hypothesis because the number of patients included in those studies is too low. The aim of the study is to compare thrombolytic treatment with heparin (which is the reference therapy for pulmonary embolism) in a large group of patients with sub-massive pulmonary embolism.

DETAILED DESCRIPTION:
A prospective, randomized, double-blind, placebo-controlled, international, multicentre, parallel-group comparison trial evaluating the efficacy and safety of single i.v. bolus tenecteplase plus standard anticoagulation as compared with standard anticoagulation in normotensive patients with acute pulmonary embolism and with echocardiographic and laboratory evidence of right ventricular dysfunction.Patients suffering from acute pulmonary embolism (first symptoms occurring within 15 days) confirmed by lung scanning or a positive spiral computed tomogram, or a positive pulmonary angiogram, presenting with right ventricular dysfunction on echocardiography and tested troponin I or T positive will be included in the study if they have no exclusion criteria.Patients in the investigational group will receive: Ø Tenecteplase as a single body-weight (known or estimated) adjusted IV bolus administered over 5 - 10 seconds not later than 30 minutes after randomization, and not later than 2 hours after the diagnosis of RV dysfunction Weight (kg) Dose in mg Dose in units Dose in ml<60 30 mg 6000 U 6 ml>60 to <70 35 mg 7000 U 7 ml>70 to <80 40 mg 8000 U 8 ml>80 to <90 45 mg 9000 U 9 ml>90 50 mg 10000 U 10 mlØ and: concomitant therapy-Unfractionated heparin at a dose of 80 IUxKg-1 as an intravenous bolus, followed by an infusion of 18 IUxKg-1xh-1, to be administered immediately after randomization in all patients for at least 48 hours following randomization. Beyond this period, intravenous UFH may be substituted with subcutaneous heparin (LMWH) treatment. The bolus will be omitted when heparin was started before randomisation.Patients in the control group will receive Ø placebo as a single body-weight (known or estimated) adjusted IV bolus administered over 5 - 10 seconds not later than 30 minutes after randomization, and not later than 2 hours after the diagnosis of RV dysfunction. Weight (kg) Dose in ml<60 6 ml>60 to <70 7 ml>70 to <80 8 ml>80 to <90 9 ml>90 10 mlØ and concomitant therapy with Unfractionated heparin

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Acute PE (first symptoms occurring 15 days or less before randomisation) confirmed by lung scan, or a positive spiral computed tomogram, or a positive pulmonary angiogram
* Right ventricular dysfunction confirmed by echocardiography or spiral computed tomography of the chest and a positive troponin I or T test

Exclusion criteria:

* Haemodynamic collapse at presentation as defined above
* Known significant bleeding risk
* Administration of thrombolytic agents within the previous 4 days
* Vena cava filter insertion or pulmonary thrombectomy within the previous 4 days
* Uncontrolled hypertension defined as systolic BP >180 mm Hg and/or diastolic BP >110 mm Hg at randomisation
* Treatment with an investigational drug under another study protocol in the previous 7 days or greater, according to local requirements
* Previous enrolment in this study
* Known hypersensitivity to tenecteplase, alteplase, unfractionated heparin, or to any of the excipients
* Pregnancy, lactation or parturition within the previous 30 days. Women of childbearing age must have a negative pregnancy test or use a medically accepted method of birth control
* Known coagulation disorder (including vitamin K antagonists)
* Any other condition that the investigator feels would place the patient at increased risk if the investigational therapy is initiated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1005 (Actual)
Dates: Start 2007-11-16 (Actual); Primary Completion 2012-07-26 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Clinical composite endpoint of all-cause mortality or haemodynamic collapse within 7 days | Day 7
Haemodynamic collapse is defined as: need for cardiopulmonary resuscitation; or systolic blood pressure < 90 mm Hg for at least 15 min or drop of syst | Day 7

SECONDARY OUTCOMES:
Death within 7 days | Day 7
Haemodynamic collapse within 7 days | Day 7
Confirmed symptomatic pulmonary embolism recurrence within 7 days | Day 7
Death within 30 days | Day 30
Total strokes (intra cranial haemorrhage or ischaemic stroke) within 7 days | Day 7
Major bleeding (other intracranial haemorrhage or ischaemic stroke) | Day 7

CONTACTS AND LOCATIONS:
Overall Officials: Guy MEYER, MD PhD, Principal Investigator — Assistance Publique Hopitaux de Paris - Department of pneumology - European Hospital George Pompidou - Paris 15; Stavros Konstantinides, MD, PhD, Principal Investigator — Department of Cardiology and Pulmonolog - Universitaetsmedizin Goettingen - 37099 Goettingen, Germany
Locations (12):
- Vienna Medical University, Vienna, Austria
- Hospital St. Luc, Brussels, Belgium
- CHU Hopital Jean Minjoz, Besançon, France
- Universistaetsklinik, Freiburg im Breisgau, Germany
- Democritus University of Thrace, Alexandroupoli, Greece
- University of Pécs, Pécs, Hungary
- Rambam Health Care Campus, Haifa, Israel
- Istituto di Cardiologia, Policlinico S.Orsola-MaBologna, Bologna, Italy
- Medical University of Warsaw, Warsaw, Poland
- Hospital Garcia de Orta, Almada, Portugal
- University Medical Center, Ljubljana, Slovenia
- Ramon y Cajal Hospital, Madrid, Spain

REFERENCES:
- [Result] Wan S, Quinlan DJ, Agnelli G, Eikelboom JW. Thrombolysis compared with heparin for the initial treatment of pulmonary embolism: a meta-analysis of the randomized controlled trials. Circulation. 2004 Aug 10;110(6):744-9. doi: 10.1161/01.CIR.0000137826.09715.9C. Epub 2004 Jul 19. PMID 15262836
- [Derived] Zuo Z, Yue J, Dong BR, Wu T, Liu GJ, Hao Q. Thrombolytic therapy for pulmonary embolism. Cochrane Database Syst Rev. 2021 Apr 15;4(4):CD004437. doi: 10.1002/14651858.CD004437.pub6. PMID 33857326
- [Derived] Konstantinides SV, Vicaut E, Danays T, Becattini C, Bertoletti L, Beyer-Westendorf J, Bouvaist H, Couturaud F, Dellas C, Duerschmied D, Empen K, Ferrari E, Galie N, Jimenez D, Kostrubiec M, Kozak M, Kupatt C, Lang IM, Lankeit M, Meneveau N, Palazzini M, Pruszczyk P, Rugolotto M, Salvi A, Sanchez O, Schellong S, Sobkowicz B, Meyer G. Impact of Thrombolytic Therapy on the Long-Term Outcome of Intermediate-Risk Pulmonary Embolism. J Am Coll Cardiol. 2017 Mar 28;69(12):1536-1544. doi: 10.1016/j.jacc.2016.12.039. PMID 28335835
- [Derived] Meyer G, Vicaut E, Danays T, Agnelli G, Becattini C, Beyer-Westendorf J, Bluhmki E, Bouvaist H, Brenner B, Couturaud F, Dellas C, Empen K, Franca A, Galie N, Geibel A, Goldhaber SZ, Jimenez D, Kozak M, Kupatt C, Kucher N, Lang IM, Lankeit M, Meneveau N, Pacouret G, Palazzini M, Petris A, Pruszczyk P, Rugolotto M, Salvi A, Schellong S, Sebbane M, Sobkowicz B, Stefanovic BS, Thiele H, Torbicki A, Verschuren F, Konstantinides SV; PEITHO Investigators. Fibrinolysis for patients with intermediate-risk pulmonary embolism. N Engl J Med. 2014 Apr 10;370(15):1402-11. doi: 10.1056/NEJMoa1302097. PMID 24716681
- [Derived] Steering Committee. Single-bolus tenecteplase plus heparin compared with heparin alone for normotensive patients with acute pulmonary embolism who have evidence of right ventricular dysfunction and myocardial injury: rationale and design of the Pulmonary Embolism Thrombolysis (PEITHO) trial. Am Heart J. 2012 Jan;163(1):33-38.e1. doi: 10.1016/j.ahj.2011.10.003. PMID 22172434